CLINICAL TRIAL: NCT05561673
Title: A Phase I/IIa, Open-label, Randomised, Controlled, Multi-country, Dose-escalation Study to Assess the Safety and Immunogenicity of AS37 in Combination With the Hepatitis B Surface Antigen (HBsAg), According to a 0-1 Month Schedule, in Healthy, HBs naïve, Adults Aged 18-45 Years
Brief Title: A Study on the Safety and Immune Response of AS37 Together With Hepatitis B Antigen in Adults Aged 18-45 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 215301; 2021-005629-25 (EudraCT Number)
Record Dates: First submitted 2022-09-28; First posted 2022-09-30 (Actual); Results first posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Hepatitis B virus; Hepatitis B surface antigen; Aluminum hydroxide; Adjuvant System; Safety; Immunogenicity
MeSH Terms: conditions — Hepatitis B | interventions — Aluminum Hydroxide; Engerix-B; Fendrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- HBs-alum Group (Active Comparator): Participants received 3 doses of GSK's Hepatitis B (HBsAg) vaccine adjuvanted with aluminum hydroxide, at Day 1, Day 31 and Day 181.
  Interventions: Combination Product: GSK's Hepatitis B vaccine adjuvanted with aluminum hydroxide
- HBs-AS03 Group (Experimental): Participants received 2 doses of GSK's HBsAg candidate vaccine adjuvanted with GSK's AS03, adjuvant system, at Day 1 and Day 31.
  Interventions: Biological: GSK's HBsAg candidate vaccine adjuvanted with GSK's AS03 adjuvant system
- HBs-AS04 Group (Experimental): Participants received 2 doses of GSK's HBsAg vaccine adjuvanted with GSK's AS04, adjuvant system, at Day 1 and Day 31.
  Interventions: Biological: GSK's Hepatitis B vaccine adjuvanted with GSK's AS04 adjuvant system
- HBs-AS37B Group (Experimental): Participants received 2 doses of GSK's HBsAg (20 µg) candidate vaccine adjuvanted with GSK's AS37B adjuvant system (50 µg), at Day 1 and Day 31.
  Interventions: Biological: GSK's HBsAg (20 μg) vaccine adjuvanted with GSK's AS37B adjuvant system (50 μg)
- HBs-AS37A Group (Experimental): Participants received 2 doses of GSK's HBsAg (20 µg) candidate vaccine adjuvanted with GSK's AS37A adjuvant system (100 µg), at Day 1 and Day 31.
  Interventions: Biological: GSK's HBsAg (20 μg) vaccine adjuvanted with GSK's AS37A adjuvant system (100 μg)

INTERVENTIONS:
Combination Product: GSK's Hepatitis B vaccine adjuvanted with aluminum hydroxide — Three doses of GSK's Hepatitis B vaccine adjuvanted with aluminum hydroxide administered intramuscularly in the non-dominant arm, one each at Day 1, Day 31 and Day 181.
  Other Names: Engerix-B
  Arms: HBs-alum Group
Biological: GSK's HBsAg candidate vaccine adjuvanted with GSK's AS03 adjuvant system — Two doses of GSK's HBsAg candidate vaccine adjuvanted with GSK's AS03 adjuvant system administered intramuscularly in the non-dominant arm, one each at Day 1 and Day 31.
  Arms: HBs-AS03 Group
Biological: GSK's Hepatitis B vaccine adjuvanted with GSK's AS04 adjuvant system — Two doses of GSK's Hepatitis B vaccine adjuvanted with GSK's AS04 adjuvant system administered intramuscularly in the non-dominant arm, one each at Day 1 and Day 31.
  Other Names: Fendrix
  Arms: HBs-AS04 Group
Biological: GSK's HBsAg (20 μg) vaccine adjuvanted with GSK's AS37B adjuvant system (50 μg) — Two doses of GSK's HBsAg (20 μg) vaccine adjuvanted with GSK's AS37B adjuvant system (50 μg) administered intramuscularly in the non-dominant arm, one each at Day 1 and Day 31.
  Arms: HBs-AS37B Group
Biological: GSK's HBsAg (20 μg) vaccine adjuvanted with GSK's AS37A adjuvant system (100 μg) — Two doses of GSK's HBsAg (20 μg )vaccine adjuvanted with GSK's AS37A adjuvant system (100 μg) administered intramuscularly in the non-dominant arm, one each at Day 1 and Day 31.
  Arms: HBs-AS37A Group

SUMMARY:
This study is conducted to assess safety and immunogenicity of GSK's HBsAg vaccine adjuvanted with GSK's AS37 adjuvant system in healthy, HBs naïve, adults aged 18-45 years and to differentiate GSK's AS37 adjuvant system from other approved adjuvant systems and from an aluminum-based adjuvant.

ELIGIBILITY:
Inclusion Criteria:

* Participants who the investigator believe can and will comply with the requirements of the protocol.
* Written informed consent obtained from the participant prior to performance of any study-specific procedure.
* Healthy participants as established by medical history, clinical examination and clinical laboratory assessment before entering the study.
* A male or female between, and including, 18 and 45 years at the time of the first study intervention administration.
* Female participants of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as pre-menarche, current bilateral tubal ligation or occlusion, hysterectomy, bilateral ovariectomy or post-menopause.
* Female participants of childbearing potential may be enrolled in the study, if the participant:

  * has practiced adequate contraception for 1 month prior to study intervention administration, and
  * has a negative pregnancy test on the day of study intervention administration, and
  * has agreed to continue adequate contraception during the entire treatment period and for at least 3 months after completion of the study intervention administration series.
  * blood sample for simultaneous follicle-stimulating hormone (FSH) and estradiol levels may be collected at the discretion of the investigator to confirm non-reproductive potential according to local laboratory reference range.

Exclusion Criteria:

Medical conditions

* Previous vaccination against Hepatitis B.
* Positive for anti-HBs antibodies or anti-HBc antibodies or HBsAg.
* Any previous administration of monophosphoryl lipid (MPL) and/or AS37.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Any confirmed or suspected autoimmune disease.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study intervention(s).
* Recurrent history or uncontrolled neurological disorders or seizures.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.
* Any clinically significant* haematological and/or biochemical laboratory abnormality.

  *The investigator should use his/her clinical judgement to decide which abnormalities are clinically significant.
* Any past or current malignancies and lymphoproliferative disorders.

Prior/Concomitant therapy

* Use of any investigational or non-registered product (drug or vaccine) other than the study intervention(s) during the period beginning 30 days before the first dose of study intervention(s) or their planned use during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before each dose and ending 30 days after each dose of study intervention(s) administration with the exception of influenza vaccine (pandemic or seasonal).
* A vaccine not foreseen by the study protocol administered during the period starting at Visit 1 or 30 days before each dose and ending 30 days after the last dose of study intervention(s) administration*, with the exception of influenza vaccine (pandemic or seasonal).

  *In case emergency mass vaccination for an unforeseen public health threat (e.g. a pandemic) is organised by public health authorities outside the routine immunisation programme, the time period described above can be reduced if necessary for that vaccine, provided it is licensed/authorised and used according to its Product Information.
* Administration of long-acting immune-modifying drugs at any time during the study period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 3 months before the first study intervention dose(s). For corticosteroids, this will mean prednisone equivalent ≥ 20 mg/day. Inhaled and topical steroids are allowed.
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 3 months before the administration of the first dose of study intervention(s) or planned administration during the study period.

Prior/Concurrent clinical study experience

* Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational intervention.

Other exclusions

* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* History of chronic alcohol consumption and/or drug abuse.
* Any study personnel or their immediate depandants, family, or household members.

Specific exclusion for MRI-assessable subgroup participants (post-randomization procedure)

* Presence of pacemakers, metal implants and/or prostheses.
* Claustrophobia.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2024-11-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- GSK Investigational Site, Leuven, Belgium
- Germany (3):
  - GSK Investigational Site, Cologne
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Magdeburg
- GSK Investigational Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer tohttps://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HBs-alum Group | HBs-AS03 Group | HBs-AS04 Group | HBs-AS37B Group | HBs-AS37A Group
Started | 25 | 25 | 24 | 25 | 23
Completed | 24 | 23 | 23 | 24 | 23
Not Completed | 1 | 2 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 0
Not completed — Consent withdrawal, not due to (S)AE | 0 | 1 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline characteristics are presented for the Exposed set, that included participants who received at least one study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | HBs-alum Group | HBs-AS03 Group | HBs-AS04 Group | HBs-AS37B Group | HBs-AS37A Group | Total
Number analyzed (Participants) | 25 | 25 | 24 | 25 | 23 | 122
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 35.9 (5.8) | 37.5 (6.4) | 34.5 (7.9) | 38.6 (6.0) | 37.3 (7.7) | 36.8 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 10 | 10 | 10 | 51
  Male | 14 | 15 | 14 | 15 | 13 | 71
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Asian and Black or African American are considered minority races in this study and are presented together under the category "Other Races".
  Participants
    Other Races | 2 | 0 | 2 | 2 | 1 | 7
    White | 23 | 25 | 22 | 23 | 22 | 115

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Administration Site Adverse Events (AEs) After Dose 1
Description: Assessed solicited administration site events after vaccination included erythema, pain, and swelling at the injection site. Any = occurrence of the event regardless of intensity grade.
Time Frame: Day 1 (day of administration) to Day 14
Population: The analysis was performed on the Exposed Set (ES), which included all participants who received at least 1 dose of the study intervention. Only participants with solicited administration site events diary card available after dose 1 administration for the specified duration were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | HBs-alum Group | HBs-AS03 Group | HBs-AS04 Group | HBs-AS37B Group | HBs-AS37A Group
Number analyzed (Participants) | 25 | 25 | 24 | 25 | 23
Participants
  Erythema | 0 | 0 | 0 | 0 | 0
  Pain | 6 | 17 | 21 | 16 | 18
  Swelling | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Solicited Administration Site AEs After Dose 2
Description: Assessed solicited administration site events after vaccination included erythema, pain and swelling at the injection site. Any = occurrence of the event regardless of intensity grade.
Time Frame: Day 31 (day of administration) to Day 45
Population: The analysis was performed on the ES. Only participants with solicited administration site events diary card available after dose 2 administration for the specified duration were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | HBs-alum Group | HBs-AS03 Group | HBs-AS04 Group | HBs-AS37B Group | HBs-AS37A Group
Number analyzed (Participants) | 24 | 24 | 23 | 25 | 23
Participants
  Erythema | 0 | 0 | 0 | 0 | 0
  Pain | 1 | 15 | 16 | 14 | 14
  Swelling | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Solicited Systemic AEs After Dose 1
Description: Assessed solicited systemic events included fever (defined as temperature greater than or equal to (>=) 38.0°C regardless of the location of measurement), fatigue, myalgia, arthralgia, headache, chills, malaise, loss of appetite, nausea, vomiting, and diarrhea.
Time Frame: Day 1 (day of administration) to Day 14
Population: The analysis was performed on the ES. Only participants with solicited systemic events diary card available after dose 1 administration for the specified duration were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | HBs-alum Group | HBs-AS03 Group | HBs-AS04 Group | HBs-AS37B Group | HBs-AS37A Group
Number analyzed (Participants) | 25 | 25 | 24 | 25 | 23
Participants
  Arthralgia | 1 | 2 | 2 | 2 | 1
  Chills | 2 | 0 | 0 | 1 | 1
  Diarrhea | 3 | 2 | 4 | 0 | 2
  Fatigue | 9 | 10 | 10 | 12 | 11
  Headache | 8 | 9 | 8 | 10 | 10
  Loss of appetite | 1 | 4 | 2 | 1 | 0
  Malaise | 8 | 2 | 7 | 3 | 2
  Myalgia | 8 | 6 | 14 | 7 | 9
  Nausea | 6 | 0 | 3 | 1 | 1
  Fever | 1 | 2 | 1 | 2 | 0
  Vomiting | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Solicited Systemic AEs After Dose 2
Description: Assessed solicited systemic events included fever (defined as temperature >=38.0°C regardless of the location of measurement), fatigue, myalgia, arthralgia, headache, chills, malaise, loss of appetite, nausea, vomiting, and diarrhea.
Time Frame: Day 31 (day of administration) to Day 45
Population: The analysis was performed on the ES. Only participants with solicited systemic events diary card available after dose 2 administration for the specified duration were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | HBs-alum Group | HBs-AS03 Group | HBs-AS04 Group | HBs-AS37B Group | HBs-AS37A Group
Number analyzed (Participants) | 24 | 24 | 23 | 25 | 23
Participants
  Arthralgia | 2 | 3 | 1 | 1 | 1
  Chills | 2 | 4 | 0 | 1 | 2
  Diarrhea | 3 | 2 | 1 | 1 | 1
  Fatigue | 9 | 8 | 8 | 7 | 5
  Headache | 9 | 8 | 7 | 7 | 4
  Loss of appetite | 3 | 2 | 0 | 0 | 1
  Malaise | 6 | 7 | 1 | 3 | 2
  Myalgia | 2 | 7 | 12 | 6 | 7
  Nausea | 2 | 1 | 3 | 1 | 2
  Fever | 1 | 1 | 1 | 1 | 1
  Vomiting | 0 | 0 | 0 | 1 | 1

5. Primary Outcome: Duration in Days of Solicited Administration Site AEs After Dose 1
Description: Duration is the number of days in which a participant experienced the symptom within the 14-day solicited follow-up period.
Time Frame: Day 1 (day of administration) to Day 14
Population: The analysis was performed on the ES. Only participants who experienced solicited administration site events after dose 1 administration for the specified duration were included in this analysis. Here, 'Number of Participants Analyzed' = participants with available data for solicited administration site events at dose 1.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | HBs-alum Group | HBs-AS03 Group | HBs-AS04 Group | HBs-AS37B Group | HBs-AS37A Group
Number analyzed (Participants) | 6 | 17 | 21 | 16 | 18
Days | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 3.0] | 3.0 [1.0 to 4.0] | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0]

6. Primary Outcome: Duration in Days of Solicited Administration Site AEs After Dose 2
Description: as for outcome 5
Time Frame: Day 31 (day of administration) to Day 45
Population: The analysis was performed on the ES. Only participants who experienced solicited administration site events after dose 2 administration for the specified duration were included in this analysis. Here, 'Number of Participants Analyzed' = participants with available data for solicited administration site events at dose 2.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | HBs-alum Group | HBs-AS03 Group | HBs-AS04 Group | HBs-AS37B Group | HBs-AS37A Group
Number analyzed (Participants) | 1 | 15 | 16 | 14 | 14
Days | 1.0 [1.0 to 1.0] | 2.0 [2.0 to 3.0] | 4.0 [2.5 to 5.0] | 1.5 [1.0 to 3.0] | 2.0 [1.0 to 3.0]

7. Primary Outcome: Duration in Days of Solicited Systemic AEs After Dose 1
Description: as for outcome 5
Time Frame: Day 1 (day of administration) to Day 14
Population: The analysis was performed on the ES. Only participants who experienced solicited systemic events after dose 1 administration for the specified duration were included in this analysis. Here, 'Number of Participants Analyzed' = participants with available data for solicited systemic events at dose 1.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | HBs-alum Group | HBs-AS03 Group | HBs-AS04 Group | HBs-AS37B Group | HBs-AS37A Group
Number analyzed (Participants) | 9 | 10 | 14 | 12 | 11
Days
  Arthralgia: number analyzed (Participants) | 1 | 2 | 2 | 2 | 1
  Arthralgia | 2.0 [2.0 to 2.0] | 1.5 [1.0 to 2.0] | 1.0 [1.0 to 1.0] | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 1.0]
  Chills: number analyzed (Participants) | 2 | 0 | 0 | 1 | 1
  Chills | 1.5 [1.0 to 2.0] |  |  | 1.0 [1.0 to 1.0] | 3.0 [3.0 to 3.0]
  Diarrhea: number analyzed (Participants) | 3 | 2 | 4 | 0 | 2
  Diarrhea | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 1.0] | 1.5 [1.0 to 2.0] |  | 1.0 [1.0 to 1.0]
  Fatigue: number analyzed (Participants) | 9 | 10 | 10 | 12 | 11
  Fatigue | 1.0 [1.0 to 3.0] | 2.0 [1.0 to 4.0] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0]
  Headache: number analyzed (Participants) | 8 | 9 | 8 | 10 | 10
  Headache | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 1.5 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 1.0]
  Loss of appetite: number analyzed (Participants) | 1 | 4 | 2 | 1 | 0
  Loss of appetite | 5.0 [5.0 to 5.0] | 1.5 [1.0 to 2.0] | 1.5 [1.0 to 2.0] | 4.0 [4.0 to 4.0] |
  Malaise: number analyzed (Participants) | 8 | 2 | 7 | 3 | 2
  Malaise | 1.0 [1.0 to 2.0] | 1.5 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 1.0]
  Myalgia: number analyzed (Participants) | 8 | 6 | 14 | 7 | 9
  Myalgia | 1.5 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 4.0] | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0]
  Nausea: number analyzed (Participants) | 6 | 0 | 3 | 1 | 1
  Nausea | 1.0 [1.0 to 2.0] |  | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  Fever: number analyzed (Participants) | 1 | 2 | 1 | 2 | 0
  Fever | 1.0 [1.0 to 1.0] | 2.5 [2.0 to 3.0] | 3.0 [3.0 to 3.0] | 3.0 [2.0 to 4.0] |

8. Primary Outcome: Duration in Days of Solicited Systemic AEs After Dose 2
Description: as for outcome 5
Time Frame: Day 31 (day of administration) to Day 45
Population: The analysis was performed on the ES. Only participants who experienced solicited systemic events after dose 2 administration for the specified duration were included in this analysis. Here, 'Number of Participants Analyzed' = participants with available data for solicited systemic events at dose 2.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | HBs-alum Group | HBs-AS03 Group | HBs-AS04 Group | HBs-AS37B Group | HBs-AS37A Group
Number analyzed (Participants) | 9 | 8 | 12 | 7 | 7
Days
  Arthralgia: number analyzed (Participants) | 2 | 3 | 1 | 1 | 1
  Arthralgia | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 1.0] | 5.0 [5.0 to 5.0] | 1.0 [1.0 to 1.0]
  Chills: number analyzed (Participants) | 2 | 4 | 0 | 1 | 2
  Chills | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.5] |  | 1.0 [1.0 to 1.0] | 1.5 [1.0 to 2.0]
  Diarrhea: number analyzed (Participants) | 3 | 2 | 1 | 1 | 1
  Diarrhea | 1.0 [1.0 to 2.0] | 1.5 [1.0 to 2.0] | 2.0 [2.0 to 2.0] | 2.0 [2.0 to 2.0] | 1.0 [1.0 to 1.0]
  Fatigue: number analyzed (Participants) | 9 | 8 | 8 | 7 | 5
  Fatigue | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.5] | 1.5 [1.0 to 4.0] | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 1.0]
  Headache: number analyzed (Participants) | 9 | 8 | 7 | 7 | 4
  Headache | 1.0 [1.0 to 1.0] | 1.5 [1.0 to 2.5] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 4.0] | 2.0 [1.0 to 3.5]
  Loss of appetite: number analyzed (Participants) | 3 | 2 | 0 | 0 | 1
  Loss of appetite | 1.0 [1.0 to 5.0] | 2.0 [1.0 to 3.0] |  |  | 1.0 [1.0 to 1.0]
  Malaise: number analyzed (Participants) | 6 | 7 | 1 | 3 | 2
  Malaise | 2.5 [2.0 to 3.0] | 1.0 [1.0 to 2.0] | 3.0 [3.0 to 3.0] | 2.0 [1.0 to 6.0] | 1.5 [1.0 to 2.0]
  Myalgia: number analyzed (Participants) | 2 | 7 | 12 | 6 | 7
  Myalgia | 2.5 [1.0 to 4.0] | 2.0 [1.0 to 4.0] | 2.5 [1.5 to 3.5] | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 3.0]
  Nausea: number analyzed (Participants) | 2 | 1 | 3 | 1 | 2
  Nausea | 2.5 [2.0 to 3.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 2.0 [2.0 to 2.0] | 1.0 [1.0 to 1.0]
  Fever: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Fever | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 4.0 [4.0 to 4.0] | 1.0 [1.0 to 1.0] | 2.0 [2.0 to 2.0]
  Vomiting: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1
  Vomiting |  |  |  | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]

9. Primary Outcome: Number of Participants With Any Unsolicited AEs After Dose 1
Description: An unsolicited AE is an AE that was not included in a list of solicited events using a Participant Diary. Unsolicited events must have been spontaneously communicated by a participant who has signed the informed consent. Unsolicited AEs include both serious and non-serious AEs. Any = occurrence of the event regardless of intensity grade or relation to the study vaccination.
Time Frame: Day 1 (day of administration) to Day 31
Population: The analysis was performed on the ES. Only participants with unsolicited AEs after dose 1 administration for the specified duration were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | HBs-alum Group | HBs-AS03 Group | HBs-AS04 Group | HBs-AS37B Group | HBs-AS37A Group
Number analyzed (Participants) | 25 | 25 | 24 | 25 | 23
Participants | 7 | 2 | 6 | 4 | 5

10. Primary Outcome: Number of Participants With Any Unsolicited AEs After Dose 2
Description: Any = occurrence of the event regardless of intensity grade or relation to the study vaccination.
Time Frame: Day 31 (day of administration) to Day 61
Population: The analysis was performed on the ES. Only participants with unsolicited AEs after dose 2 administration for the specified duration were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | HBs-alum Group | HBs-AS03 Group | HBs-AS04 Group | HBs-AS37B Group | HBs-AS37A Group
Number analyzed (Participants) | 24 | 24 | 23 | 25 | 23
Participants | 5 | 7 | 6 | 6 | 6

11. Primary Outcome: Number of Participants With Serious AEs (SAEs)
Description: An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant, or is an abnormal pregnancy outcome. Any = occurrence of the SAE regardless of intensity grade or relation to the study vaccination.
Time Frame: Throughout the entire study period (from Day 1 to Day 361)
Population: The analysis was performed on the ES.
Measure: Count of Participants; unit: Participants
Arm/Group | HBs-alum Group | HBs-AS03 Group | HBs-AS04 Group | HBs-AS37B Group | HBs-AS37A Group
Number analyzed (Participants) | 25 | 25 | 24 | 25 | 23
Participants | 0 | 0 | 0 | 1 | 0

12. Primary Outcome: Number of Participants With Medically Attended AEs (MAEs)
Description: An MAE is any AE with medically attended visits that were not routine visits for physical examination or vaccination, such as visits for hospitalization, an emergency room visit, or an otherwise unscheduled visit to or from medical personnel (medical doctor) for any reason. Any = occurrence of the MAE regardless of intensity grade or relation to the study vaccination.
Time Frame: Throughout the entire study period (from Day 1 to Day 361)
Population: The analysis was performed on the ES.
Measure: Count of Participants; unit: Participants
Arm/Group | HBs-alum Group | HBs-AS03 Group | HBs-AS04 Group | HBs-AS37B Group | HBs-AS37A Group
Number analyzed (Participants) | 25 | 25 | 24 | 25 | 23
Participants | 8 | 2 | 2 | 3 | 4

13. Primary Outcome: Number of Participants With AEs Leading to Study Withdrawal
Description: An AE is any untoward medical occurrence (an unfavourable/unintended sign - including an abnormal laboratory finding), symptom, or disease (new or exacerbated) in a clinical study participant that is temporally associated with the study intervention. The AE may or may not be considered related to the study intervention. A participant is considered to have withdrawn from the study if no new study procedure has been performed or no new information has been collected for him/her since the date of withdrawal/last contact.
Time Frame: Throughout the entire study period (from Day 1 to Day 361)
Population: The analysis was performed on the ES.
Measure: Count of Participants; unit: Participants
Arm/Group | HBs-alum Group | HBs-AS03 Group | HBs-AS04 Group | HBs-AS37B Group | HBs-AS37A Group
Number analyzed (Participants) | 25 | 25 | 24 | 25 | 23
Participants | 0 | 0 | 0 | 0 | 0

14. Primary Outcome: Number of Participants With Potential Mediated Immune Diseases (pIMDs)
Description: pIMDs are a subset of adverse events that include autoimmune diseases and other inflammatory and/or neurological disorders of interest which may or may not have an autoimmune aetiology. Any = occurrence of the pIMD regardless of intensity grade or relation to the study vaccination.
Time Frame: Throughout the entire study period (from Day 1 to Day 361)
Population: The analysis was performed on the ES.
Measure: Count of Participants; unit: Participants
Arm/Group | HBs-alum Group | HBs-AS03 Group | HBs-AS04 Group | HBs-AS37B Group | HBs-AS37A Group
Number analyzed (Participants) | 25 | 25 | 24 | 25 | 23
Participants | 0 | 0 | 0 | 1 | 0

15. Primary Outcome: Mean Percent Change From Baseline (Pre-vaccination, Day 1) in Hematology and Biochemistry Parameters Post-dose 1
Description: In the analysis were included biochemistry parameters: alanine aminotransferase (ALT), aspartate aminotransferase (AST), bicarbonate, blood urea nitrogen, chloride, C reactive protein, creatinine, potassium, sodium; and hematology parameters: eosinophils, erythrocytes, hemoglobin, lymphocytes, platelets, monocytes, neutrophils, white blood cells (WBC).
Time Frame: At Day 8 (relative to baseline [pre-vaccination Day 1])
Population: The analysis was performed on the ES. Only participants for whom the specified laboratory data after dose 1 administration were available for the specified timepoint (at Day 8) were included in analysis.
Measure: Mean (Standard Deviation); unit: Mean percent change from baseline
Arm/Group | HBs-alum Group | HBs-AS03 Group | HBs-AS04 Group | HBs-AS37B Group | HBs-AS37A Group
Number analyzed (Participants) | 25 | 25 | 24 | 25 | 23
Mean percent change from baseline
  ALT | -3.04 (20.322) | -6.69 (14.117) | -1.13 (34.221) | 8.14 (25.853) | 0.95 (15.926)
  AST | 4.74 (17.106) | -5.62 (14.509) | -1.79 (18.626) | 7.35 (24.486) | 2.28 (16.477)
  Bicarbonate | 0.52 (7.789) | -0.19 (8.276) | 3.68 (8.491) | 0.06 (10.180) | 4.16 (7.337)
  Blood urea nitrogen | 2.60 (29.717) | -3.03 (19.264) | 1.84 (32.456) | 0.09 (25.501) | -0.63 (15.543)
  Chloride | 0.79 (1.921) | 0.23 (2.119) | -0.11 (2.000) | -0.33 (2.247) | -0.24 (2.119)
  C Reactive Protein | 78.43 (349.570) | 41.16 (124.844) | 129.65 (393.365) | 5.72 (57.451) | -6.50 (45.671)
  Creatinine | 0.34 (8.164) | -2.35 (10.278) | -2.01 (7.209) | -0.10 (9.989) | 0.76 (9.176)
  Potassium | 1.88 (8.648) | -0.14 (8.133) | 1.91 (8.313) | 2.43 (7.932) | 0.27 (6.323)
  Sodium | 0.26 (1.204) | 0.18 (1.376) | 0.27 (1.438) | 0.04 (1.481) | 0.19 (1.253)
  Eosinophils: number analyzed (Participants) | 24 | 25 | 24 | 24 | 22
  Eosinophils | 20.35 (45.285) | 31.51 (76.423) | -3.33 (46.839) | 18.15 (45.276) | 12.86 (38.767)
  Erythrocytes: number analyzed (Participants) | 24 | 25 | 24 | 25 | 22
  Erythrocytes | -2.06 (3.756) | -1.01 (3.786) | -0.67 (4.423) | 0.45 (5.160) | -0.21 (4.384)
  Hemoglobin: number analyzed (Participants) | 24 | 25 | 24 | 25 | 22
  Hemoglobin | -2.17 (3.729) | -0.94 (3.817) | -0.60 (3.892) | 0.74 (5.156) | -0.36 (4.075)
  Lymphocytes: number analyzed (Participants) | 24 | 25 | 24 | 24 | 22
  Lymphocytes | 8.79 (18.849) | 6.58 (23.996) | 1.25 (25.224) | 7.80 (32.898) | 4.04 (15.252)
  Platelets: number analyzed (Participants) | 24 | 25 | 23 | 25 | 22
  Platelets | 1.56 (10.141) | 2.84 (7.234) | 5.10 (10.605) | 4.72 (10.952) | 5.67 (11.517)
  Monocytes: number analyzed (Participants) | 24 | 25 | 24 | 24 | 22
  Monocytes | 8.83 (23.264) | 6.20 (24.148) | 7.31 (36.121) | 12.52 (35.758) | 4.98 (24.417)
  Neutrophils: number analyzed (Participants) | 24 | 25 | 24 | 24 | 22
  Neutrophils | 2.69 (27.341) | -2.23 (28.410) | 14.24 (38.460) | 2.03 (25.842) | 4.70 (28.444)
  WBC: number analyzed (Participants) | 24 | 25 | 24 | 25 | 22
  WBC | 4.06 (16.847) | 0.88 (17.754) | 7.58 (19.074) | 0.26 (21.314) | 3.53 (18.126)

16. Primary Outcome: Mean Percent Change From Baseline (Pre-vaccination, Day 1) in Hematology and Biochemistry Parameters Post-dose 1
Description: In the analysis were included biochemistry parameters: ALT, AST, bicarbonate, blood urea nitrogen, chloride, C reactive protein, creatinine, potassium, sodium; and hematology parameters: eosinophils, erythrocytes, hemoglobin, lymphocytes, platelets, monocytes, neutrophils, WBC.
Time Frame: At Day 31 (compared with baseline [prevaccination, Day 1])
Population: The analysis was performed on the ES. Only participants for whom the specified laboratory data after dose 1 administration were available for the specified timepoint (at Day 31) were included in analysis.
Measure: Mean (Standard Deviation); unit: Mean percent change from baseline
Arm/Group | HBs-alum Group | HBs-AS03 Group | HBs-AS04 Group | HBs-AS37B Group | HBs-AS37A Group
Number analyzed (Participants) | 24 | 24 | 23 | 25 | 23
Mean percent change from baseline
  ALT: number analyzed (Participants) | 24 | 24 | 23 | 24 | 23
  ALT | -2.45 (32.837) | 12.52 (81.650) | 2.94 (25.235) | 5.89 (25.561) | 3.07 (27.915)
  AST: number analyzed (Participants) | 24 | 24 | 23 | 24 | 23
  AST | -0.60 (22.151) | 0.12 (25.394) | 3.33 (31.456) | 3.21 (22.040) | 4.57 (21.930)
  Bicarbonate: number analyzed (Participants) | 24 | 24 | 23 | 24 | 23
  Bicarbonate | 0.58 (11.020) | -2.47 (9.490) | 0.78 (10.526) | -0.20 (9.834) | 4.65 (12.535)
  Blood urea nitrogen: number analyzed (Participants) | 24 | 24 | 23 | 24 | 23
  Blood urea nitrogen | -1.04 (17.638) | 1.42 (23.387) | -5.65 (27.995) | -3.27 (27.699) | 3.70 (23.551)
  Chloride: number analyzed (Participants) | 24 | 24 | 23 | 24 | 23
  Chloride | 0.76 (2.430) | 0.29 (2.668) | -0.16 (1.836) | 0.09 (2.059) | 0.17 (2.022)
  C Reactive Protein | 23.07 (94.084) | 37.95 (143.597) | 130.90 (518.895) | 12.48 (63.081) | 77.00 (358.139)
  Creatinine: number analyzed (Participants) | 24 | 24 | 23 | 24 | 23
  Creatinine | -3.73 (8.529) | -4.69 (9.817) | -1.37 (7.374) | -1.77 (9.931) | -2.23 (9.222)
  Potassium: number analyzed (Participants) | 24 | 24 | 23 | 24 | 23
  Potassium | -1.60 (6.867) | 0.23 (7.493) | -0.78 (7.674) | 2.46 (8.750) | -1.54 (6.611)
  Sodium: number analyzed (Participants) | 24 | 24 | 23 | 24 | 23
  Sodium | 0.18 (1.273) | 0.49 (1.486) | -0.28 (1.113) | 0.31 (1.221) | 0.13 (1.318)
  Eosinophils: number analyzed (Participants) | 24 | 24 | 23 | 24 | 23
  Eosinophils | 61.95 (156.721) | 10.80 (47.476) | 6.13 (42.536) | 43.03 (99.613) | 0.88 (44.640)
  Erythrocytes: number analyzed (Participants) | 24 | 24 | 23 | 24 | 23
  Erythrocytes | -2.30 (3.813) | -0.71 (3.877) | -1.14 (5.730) | 0.76 (4.317) | -1.06 (5.496)
  Hemoglobin: number analyzed (Participants) | 24 | 24 | 23 | 24 | 23
  Hemoglobin | -1.99 (4.925) | -0.25 (3.795) | -0.75 (5.168) | 0.92 (4.328) | -1.06 (4.325)
  Lymphocytes: number analyzed (Participants) | 24 | 24 | 23 | 24 | 23
  Lymphocytes | 3.44 (15.877) | 5.02 (23.147) | 4.16 (24.245) | -0.47 (22.632) | 0.61 (17.722)
  Platelets: number analyzed (Participants) | 24 | 24 | 23 | 24 | 23
  Platelets | -4.21 (10.893) | -1.86 (13.771) | 1.72 (10.562) | 2.92 (9.752) | 0.68 (10.344)
  Monocytes: number analyzed (Participants) | 24 | 24 | 23 | 24 | 23
  Monocytes | 8.76 (44.115) | 9.84 (30.487) | 5.31 (30.151) | 7.75 (34.218) | 9.96 (29.752)
  Neutrophils: number analyzed (Participants) | 24 | 24 | 23 | 24 | 23
  Neutrophils | 10.63 (43.055) | 2.47 (29.935) | 8.26 (27.070) | -0.67 (24.740) | 12.13 (32.091)
  WBC: number analyzed (Participants) | 24 | 24 | 23 | 24 | 23
  WBC | 6.65 (26.757) | 2.37 (18.732) | 5.78 (20.170) | -2.04 (18.832) | 6.17 (19.512)

17. Primary Outcome: Mean Percent Change From Baseline (Pre-vaccination, Day 1) in Hematology and Biochemistry Parameters Post-dose 2
Description: as for outcome 16
Time Frame: At Day 38 (compared with baseline [pre-vaccination, Day 1])
Population: The analysis was performed on the ES. Only participants for whom the specified laboratory data after dose 2 administration were available for the specified timepoint (at Day 38) were included in analysis.
Measure: Mean (Standard Deviation); unit: Mean percent change from baseline
Arm/Group | HBs-alum Group | HBs-AS03 Group | HBs-AS04 Group | HBs-AS37B Group | HBs-AS37A Group
Number analyzed (Participants) | 23 | 23 | 22 | 25 | 23
Mean percent change from baseline
  ALT | -1.70 (28.091) | -9.56 (28.152) | 8.70 (40.893) | 7.81 (24.159) | -4.15 (19.568)
  AST | 1.91 (26.199) | -7.81 (21.151) | 11.34 (41.922) | 5.63 (17.430) | -2.19 (18.087)
  Bicarbonate | -0.10 (11.002) | 1.04 (7.590) | 4.41 (12.016) | 0.75 (9.389) | 5.04 (11.085)
  Blood urea nitrogen | 2.83 (30.148) | -1.73 (23.632) | 2.30 (39.154) | 0.69 (28.712) | 5.34 (23.796)
  Chloride | 0.39 (1.824) | -0.18 (2.413) | -0.96 (2.079) | -0.46 (2.004) | 0.39 (2.058)
  C Reactive Protein | 57.03 (191.211) | 131.87 (475.577) | 55.41 (110.350) | 146.04 (584.663) | 3.02 (66.364)
  Creatinine | 1.18 (10.007) | -2.71 (8.546) | -0.25 (7.389) | 0.61 (11.670) | 1.40 (9.723)
  Potassium | -0.11 (8.188) | 0.30 (10.244) | 1.76 (10.350) | 1.83 (8.246) | 2.15 (7.425)
  Sodium | 0.31 (0.802) | 0.32 (1.833) | -0.03 (1.268) | 0.01 (1.225) | 0.38 (1.128)
  Eosinophils: number analyzed (Participants) | 22 | 23 | 22 | 25 | 23
  Eosinophils | 103.21 (216.663) | 64.45 (142.771) | 27.38 (65.060) | 35.67 (96.666) | 6.21 (58.498)
  Erythrocytes | -2.59 (4.677) | -0.54 (3.879) | 0.01 (5.660) | 0.66 (4.466) | -1.46 (5.741)
  Hemoglobin | -1.89 (5.602) | -0.44 (3.530) | -0.05 (5.064) | 0.88 (4.548) | -2.32 (3.201)
  Lymphocytes: number analyzed (Participants) | 22 | 23 | 22 | 25 | 23
  Lymphocytes | 2.35 (22.056) | 8.61 (23.233) | 15.80 (31.316) | 2.46 (25.691) | 0.10 (23.742)
  Platelets | 1.41 (11.656) | 5.25 (14.869) | 6.56 (11.374) | 2.33 (10.113) | 3.02 (14.577)
  Monocytes: number analyzed (Participants) | 22 | 23 | 22 | 25 | 23
  Monocytes | 20.33 (52.053) | 5.44 (29.929) | 23.51 (31.162) | 10.00 (32.556) | 10.95 (42.691)
  Neutrophils: number analyzed (Participants) | 22 | 23 | 22 | 25 | 23
  Neutrophils | 8.11 (39.675) | 10.17 (55.015) | 12.80 (27.430) | -5.36 (24.208) | -3.26 (32.341)
  WBC | 5.34 (24.916) | 8.19 (34.765) | 12.42 (18.141) | -3.72 (16.095) | -3.79 (19.528)

18. Primary Outcome: Mean Percent Change From Baseline (Pre-vaccination, Day 1) in Hematology and Biochemistry Parameters Post-dose 2
Description: as for outcome 16
Time Frame: At Day 61 (compared with baseline [pre-vaccination, Day 1])
Population: The analysis was performed on the ES. Only participants for whom the specified laboratory data after dose 2 administration were available for the specified timepoint (at Day 61) were included in analysis.
Measure: Mean (Standard Deviation); unit: Mean percent change from baseline
Arm/Group | HBs-alum Group | HBs-AS03 Group | HBs-AS04 Group | HBs-AS37B Group | HBs-AS37A Group
Number analyzed (Participants) | 24 | 24 | 23 | 25 | 23
Mean percent change from baseline
  ALT | -4.71 (27.145) | 61.39 (318.144) | 12.94 (49.927) | 4.67 (36.939) | 13.83 (63.700)
  AST | 8.19 (43.555) | 42.91 (171.398) | 18.51 (68.383) | 8.78 (47.643) | 3.47 (33.308)
  Bicarbonate | 0.66 (8.676) | -2.36 (8.453) | 3.17 (9.880) | -3.21 (10.373) | 4.64 (12.554)
  Blood urea nitrogen | 8.26 (26.719) | -1.24 (32.101) | -4.94 (21.078) | -2.00 (25.429) | 2.60 (21.312)
  Chloride | -0.22 (2.006) | 0.48 (2.157) | 0.09 (1.691) | -0.14 (2.311) | 0.01 (1.803)
  C Reactive Protein: number analyzed (Participants) | 24 | 24 | 22 | 25 | 23
  C Reactive Protein | 64.02 (180.495) | 121.89 (432.514) | 79.61 (218.741) | 91.49 (237.304) | 109.50 (512.035)
  Creatinine | 2.96 (13.010) | -1.84 (13.034) | 1.15 (11.041) | -3.95 (8.215) | -1.20 (7.048)
  Potassium | 0.33 (9.316) | 3.34 (10.727) | -1.88 (7.115) | 1.17 (8.379) | -0.21 (6.832)
  Sodium | -0.35 (1.278) | 0.34 (1.881) | 0.44 (1.278) | -0.33 (1.156) | 0.25 (1.335)
  Eosinophils: number analyzed (Participants) | 23 | 24 | 23 | 25 | 23
  Eosinophils | 20.20 (32.608) | 32.37 (59.533) | 42.38 (91.920) | 57.74 (144.539) | 17.59 (63.368)
  Erythrocytes: number analyzed (Participants) | 23 | 24 | 23 | 25 | 23
  Erythrocytes | -0.86 (5.037) | 0.65 (5.327) | -0.76 (5.901) | 0.51 (4.813) | -0.63 (5.596)
  Hemoglobin: number analyzed (Participants) | 23 | 24 | 23 | 25 | 23
  Hemoglobin | -0.86 (6.190) | 0.49 (4.971) | -0.85 (5.363) | 0.60 (4.671) | -1.01 (3.466)
  Lymphocytes: number analyzed (Participants) | 23 | 24 | 23 | 25 | 23
  Lymphocytes | 6.43 (21.692) | 2.32 (18.547) | 9.74 (32.460) | -1.74 (27.336) | 4.92 (21.356)
  Platelets: number analyzed (Participants) | 22 | 24 | 23 | 24 | 23
  Platelets | -1.29 (11.369) | 2.12 (15.566) | 1.35 (12.342) | 3.77 (10.156) | 3.47 (11.839)
  Monocytes: number analyzed (Participants) | 23 | 24 | 23 | 25 | 23
  Monocytes | 21.95 (56.206) | 12.47 (32.131) | 15.05 (30.852) | 5.66 (35.371) | 15.01 (42.423)
  Neutrophils: number analyzed (Participants) | 23 | 24 | 23 | 25 | 23
  Neutrophils | 3.81 (33.133) | -6.10 (40.627) | 8.68 (31.904) | 4.91 (34.720) | 12.12 (42.077)
  WBC: number analyzed (Participants) | 23 | 24 | 23 | 25 | 23
  WBC | 5.16 (22.729) | -3.20 (25.520) | 9.32 (24.511) | 0.84 (24.001) | 7.14 (25.180)

19. Secondary Outcome: Geometric Mean Concentration (GMC) of Anti-HBs Antibody Concentrations
Description: Anti-HBs antibody concentration was measured as GMC and expressed in milli international units per milliliter (mIU/mL).
Time Frame: At Day 1, Day 31, Day 61 and Day 361
Population: The analysis was performed on the Per-Protocol set (PPS), which included all participants who received all doses as per protocol, had immunogenicity results post-dose, complied with dosing/blood draw intervals, without intercurrent conditions that may interfere with immunogenicity and without prohibited concomitant medication/vaccination. Only participants with data available for GMC of anti-HBs antibody concentration at the specified timepoints were included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | HBs-alum Group | HBs-AS03 Group | HBs-AS04 Group | HBs-AS37B Group | HBs-AS37A Group
Number analyzed (Participants) | 25 | 24 | 23 | 24 | 23
mIU/mL
  Day 1 | 3.4 [3.0 to 3.8] | 3.1 [3.1 to 3.1] | 3.1 [3.1 to 3.1] | 3.1 [3.1 to 3.1] | 3.1 [3.1 to 3.1]
  Day 31: number analyzed (Participants) | 24 | 22 | 23 | 22 | 21
  Day 31 | 7.7 [3.0 to 20.0] | 204.9 [62.8 to 668.4] | 8.3 [3.4 to 20.2] | 22.0 [10.4 to 46.6] | 95.2 [27.6 to 327.5]
  Day 61: number analyzed (Participants) | 24 | 21 | 23 | 22 | 21
  Day 61 | 40.3 [14.3 to 113.1] | 7193.0 [4062.5 to 12735.8] | 86.3 [41.1 to 181.0] | 401.3 [212.0 to 759.8] | 1574.2 [600.6 to 4125.7]
  Day 361: number analyzed (Participants) | 21 | 19 | 22 | 20 | 23
  Day 361 | 1055.9 [359.2 to 3103.7] | 3211.8 [2252.4 to 4579.7] | 41.4 [18.9 to 90.6] | 153.2 [81.6 to 287.7] | 586.3 [242.2 to 1419.4]

20. Secondary Outcome: Percentage of Participants Who Seroconverted for Anti-HBs
Description: A participant who seroconverted for anti-HBs is defined as a participant with an anti-HBs antibody concentration higher than (>) 6.2 mIU/mL.
Time Frame: At Day 31, Day 61 and Day 361
Population: The analysis was performed on the PPS. Only participants that seroconverted for anti-HBs and had data available at the specified timepoints were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HBs-alum Group | HBs-AS03 Group | HBs-AS04 Group | HBs-AS37B Group | HBs-AS37A Group
Number analyzed (Participants) | 24 | 22 | 23 | 22 | 23
Percentage of participants
  Day 31: number analyzed (Participants) | 24 | 22 | 23 | 22 | 21
  Day 31 | 16.7 [4.7 to 37.4] | 95.5 [77.2 to 99.9] | 21.7 [7.5 to 43.7] | 59.1 [36.4 to 79.3] | 81.0 [58.1 to 94.6]
  Day 61: number analyzed (Participants) | 24 | 21 | 23 | 22 | 21
  Day 61 | 75.0 [53.3 to 90.2] | 100 [83.9 to 100] | 87.0 [66.4 to 97.2] | 100 [84.6 to 100] | 100 [83.9 to 100]
  Day 361: number analyzed (Participants) | 21 | 19 | 22 | 20 | 23
  Day 361 | 95.2 [76.2 to 99.9] | 100 [82.4 to 100] | 72.7 [49.8 to 89.3] | 100 [83.2 to 100] | 100 [85.2 to 100]

21. Secondary Outcome: Percentage of Participants Seroprotected for Anti-HBs
Description: A participant seroprotected for anti-HBs is defined as a participant with an anti-HBs antibody concentration >10 mIU/mL.
Time Frame: At Day 31, Day 61 and Day 361
Population: The analysis was performed on the PPS. Only participants that were seroprotected for anti-HBs and had data available at the specified timepoints were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HBs-alum Group | HBs-AS03 Group | HBs-AS04 Group | HBs-AS37B Group | HBs-AS37A Group
Number analyzed (Participants) | 24 | 22 | 23 | 22 | 23
Percentage of participants
  Day 31: number analyzed (Participants) | 24 | 22 | 23 | 22 | 21
  Day 31 | 16.7 [4.7 to 37.4] | 95.5 [77.2 to 99.9] | 21.7 [7.5 to 43.7] | 59.1 [36.4 to 79.3] | 81.0 [58.1 to 94.6]
  Day 61: number analyzed (Participants) | 24 | 21 | 23 | 22 | 21
  Day 61 | 62.5 [40.6 to 81.2] | 100 [83.9 to 100] | 87.0 [66.4 to 97.2] | 100 [84.6 to 100] | 100 [83.9 to 100]
  Day 361: number analyzed (Participants) | 21 | 19 | 22 | 20 | 23
  Day 361 | 95.2 [76.2 to 99.9] | 100 [82.4 to 100] | 72.7 [49.8 to 89.3] | 100 [83.2 to 100] | 100 [85.2 to 100]

22. Primary Outcome: Number of Participants With Abnormal Hematology and Biochemistry Laboratory Parameter Values at Day 1
Description: In the analysis were included biochemistry parameters: ALT, AST, bicarbonate, blood urea nitrogen, chloride, C reactive protein, creatinine, potassium, sodium; and hematology parameters: eosinophils, erythrocytes, hemoglobin, lymphocytes, platelets, monocytes, neutrophils, WBC. Below = value below the laboratory reference range defined for the specified visit and laboratory parameter; Within = value within the laboratory reference range defined for the specified visit and laboratory parameter; Above = value above the laboratory reference range defined for the specified visit and laboratory parameter.
Time Frame: At Day 1 (baseline)
Population: The analysis was performed on the ES. Only participants for whom the specified laboratory data were available for the specified timepoint (Day 1) were included in analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | HBs-alum Group | HBs-AS03 Group | HBs-AS04 Group | HBs-AS37B Group | HBs-AS37A Group
Number analyzed (Participants) | 25 | 25 | 24 | 25 | 23
Participants
  ALT: Below | 0 | 0 | 0 | 0 | 0
  ALT: Within | 21 | 21 | 23 | 23 | 21
  ALT: Above | 4 | 4 | 1 | 2 | 2
  ALT: Missing | 0 | 0 | 0 | 0 | 0
  AST: Below | 0 | 0 | 0 | 0 | 0
  AST: Within | 22 | 24 | 24 | 25 | 22
  AST: Above | 3 | 1 | 0 | 0 | 1
  AST: Missing | 0 | 0 | 0 | 0 | 0
  Bicarbonate, Day 1: Below | 0 | 0 | 0 | 0 | 1
  Bicarbonate, Day 1: Within | 25 | 25 | 24 | 25 | 22
  Bicarbonate, Day 1: Above | 0 | 0 | 0 | 0 | 0
  Bicarbonate, Day 1: Missing | 0 | 0 | 0 | 0 | 0
  Blood urea nitrogen: Below | 0 | 0 | 0 | 0 | 0
  Blood urea nitrogen: Within | 24 | 23 | 22 | 24 | 23
  Blood urea nitrogen: Above | 1 | 2 | 2 | 1 | 0
  Blood urea nitrogen: Missing | 0 | 0 | 0 | 0 | 0
  Chloride: Below | 0 | 0 | 0 | 0 | 0
  Chloride: Within | 25 | 24 | 24 | 25 | 23
  Chloride: Above | 0 | 1 | 0 | 0 | 0
  Chloride: Missing | 0 | 0 | 0 | 0 | 0
  C Reactive Protein: Below | 0 | 0 | 0 | 0 | 0
  C Reactive Protein: Within | 24 | 24 | 21 | 23 | 20
  C Reactive Protein: Above | 1 | 1 | 3 | 2 | 3
  C Reactive Protein: Missing | 0 | 0 | 0 | 0 | 0
  Creatinine: Below | 0 | 0 | 0 | 0 | 0
  Creatinine: Within | 24 | 22 | 22 | 23 | 23
  Creatinine: Above | 1 | 3 | 2 | 2 | 0
  Creatinine: Missing | 0 | 0 | 0 | 0 | 0
  Potassium: Below | 0 | 0 | 1 | 0 | 0
  Potassium: Within | 25 | 25 | 23 | 25 | 23
  Potassium: Above | 0 | 0 | 0 | 0 | 0
  Potassium: Missing | 0 | 0 | 0 | 0 | 0
  Sodium: Below | 0 | 0 | 0 | 1 | 0
  Sodium: Within | 25 | 25 | 24 | 24 | 23
  Sodium: Above | 0 | 0 | 0 | 0 | 0
  Sodium: Missing | 0 | 0 | 0 | 0 | 0
  Eosinophils: Below | 1 | 1 | 1 | 3 | 2
  Eosinophils: Within | 24 | 23 | 22 | 21 | 21
  Eosinophils: Above | 0 | 1 | 1 | 1 | 0
  Eosinophils: Missing | 0 | 0 | 0 | 0 | 0
  Erythrocytes: Below | 1 | 1 | 3 | 2 | 1
  Erythrocytes: Within | 24 | 24 | 21 | 22 | 22
  Erythrocytes: Above | 0 | 0 | 0 | 1 | 0
  Erythrocytes: Missing | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Below | 3 | 0 | 5 | 3 | 3
  Hemoglobin: Within | 22 | 25 | 19 | 22 | 20
  Hemoglobin: Above | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Missing | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Below | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Within | 25 | 25 | 24 | 25 | 23
  Lymphocytes: Above | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Missing | 0 | 0 | 0 | 0 | 0
  Platelets: Below | 0 | 0 | 0 | 0 | 0
  Platelets: Within | 25 | 24 | 22 | 25 | 23
  Platelets: Above | 0 | 1 | 2 | 0 | 0
  Platelets: Missing | 0 | 0 | 0 | 0 | 0
  Monocytes: Below | 0 | 0 | 0 | 0 | 1
  Monocytes: Within | 25 | 25 | 24 | 25 | 22
  Monocytes: Above | 0 | 0 | 0 | 0 | 0
  Monocytes: Missing | 0 | 0 | 0 | 0 | 0
  Neutrophils: Below | 1 | 1 | 2 | 1 | 1
  Neutrophils: Within | 24 | 24 | 22 | 24 | 22
  Neutrophils: Above | 0 | 0 | 0 | 0 | 0
  Neutrophils: Missing | 0 | 0 | 0 | 0 | 0
  WBC: number analyzed (Participants) | 24 | 25 | 24 | 25 | 23
  WBC: Below | 3 | 1 | 1 | 0 | 1
  WBC: Within | 21 | 23 | 23 | 24 | 22
  WBC: Above | 0 | 1 | 0 | 1 | 0
  WBC: Missing | 0 | 0 | 0 | 0 | 0

23. Primary Outcome: Number of Participants With Abnormal Hematology and Biochemistry Laboratory Parameter Values at Day 8
Description: In the analysis were included biochemistry parameters: alanine aminotransferase (ALT), aspartate transaminase (AST), bicarbonate, blood urea nitrogen, chloride, C reactive protein, creatinine, potassium, sodium; and hematology parameters: eosinophils, erythrocytes, hemoglobin, lymphocytes, platelets, monocytes, neutrophils, white blood cells (WBC).Below = value below the laboratory reference range defined for the specified visit and laboratory parameter; Within = value within the laboratory reference range defined for the specified visit and laboratory parameter; Above = value above the laboratory reference range defined for the specified visit and laboratory parameter.
Time Frame: At Day 8
Population: The analysis was performed on the ES. Only participants for whom the specified laboratory data were available for the specified timepoint (Day 8) were included in analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | HBs-alum Group | HBs-AS03 Group | HBs-AS04 Group | HBs-AS37B Group | HBs-AS37A Group
Number analyzed (Participants) | 25 | 25 | 24 | 25 | 23
Participants
  ALT: Below | 0 | 0 | 0 | 0 | 0
  ALT: Within | 23 | 22 | 22 | 22 | 21
  ALT: Above | 2 | 3 | 2 | 3 | 2
  ALT: Missing | 0 | 0 | 0 | 0 | 0
  AST: Below | 0 | 0 | 0 | 0 | 0
  AST: Within | 24 | 24 | 24 | 24 | 23
  AST: Above | 1 | 1 | 0 | 1 | 0
  AST: Missing | 0 | 0 | 0 | 0 | 0
  Bicarbonate: Below | 0 | 0 | 0 | 0 | 0
  Bicarbonate: Within | 24 | 25 | 24 | 25 | 23
  Bicarbonate: Above | 1 | 0 | 0 | 0 | 0
  Bicarbonate: Missing | 0 | 0 | 0 | 0 | 0
  Blood urea nitrogen: Below | 0 | 0 | 0 | 0 | 0
  Blood urea nitrogen: Within | 25 | 22 | 23 | 25 | 22
  Blood urea nitrogen: Above | 0 | 3 | 1 | 0 | 1
  Blood urea nitrogen: Missing | 0 | 0 | 0 | 0 | 0
  Chloride: Below | 0 | 0 | 0 | 0 | 1
  Chloride: Within | 25 | 25 | 23 | 25 | 22
  Chloride: Above | 0 | 0 | 1 | 0 | 0
  Chloride: Missing | 0 | 0 | 0 | 0 | 0
  C Reactive Protein: Below | 0 | 0 | 0 | 0 | 0
  C Reactive Protein: Within | 23 | 24 | 21 | 24 | 21
  C Reactive Protein: Above | 2 | 1 | 3 | 1 | 2
  C Reactive Protein: Missing | 0 | 0 | 0 | 0 | 0
  Creatinine: Below | 0 | 0 | 0 | 0 | 0
  Creatinine: Within | 23 | 23 | 24 | 24 | 20
  Creatinine: Above | 2 | 2 | 0 | 1 | 3
  Creatinine: Missing | 0 | 0 | 0 | 0 | 0
  Potassium: Below | 0 | 0 | 0 | 0 | 0
  Potassium: Within | 24 | 25 | 23 | 24 | 23
  Potassium: Above | 1 | 0 | 1 | 1 | 0
  Potassium: Missing | 0 | 0 | 0 | 0 | 0
  Sodium: Below | 0 | 0 | 0 | 0 | 1
  Sodium: Within | 25 | 25 | 24 | 25 | 22
  Sodium: Above | 0 | 0 | 0 | 0 | 0
  Sodium: Missing | 0 | 0 | 0 | 0 | 0
  Eosinophils: Below | 2 | 0 | 1 | 2 | 2
  Eosinophils: Within | 22 | 24 | 23 | 21 | 19
  Eosinophils: Above | 0 | 1 | 0 | 1 | 1
  Eosinophils: Missing | 1 | 0 | 0 | 1 | 1
  Erythrocytes: Below | 1 | 0 | 2 | 1 | 1
  Erythrocytes: Within | 23 | 25 | 22 | 23 | 21
  Erythrocytes: Above | 0 | 0 | 0 | 1 | 0
  Erythrocytes: Missing | 1 | 0 | 0 | 0 | 1
  Hemoglobin: Below | 4 | 0 | 5 | 1 | 3
  Hemoglobin: Within | 20 | 25 | 19 | 24 | 19
  Hemoglobin: Above | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Missing | 1 | 0 | 0 | 0 | 1
  Lymphocytes: Below | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Within | 24 | 25 | 24 | 24 | 22
  Lymphocytes: Above | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Missing | 1 | 0 | 0 | 1 | 1
  Platelets: Below | 0 | 0 | 0 | 0 | 0
  Platelets: Within | 24 | 23 | 22 | 25 | 22
  Platelets: Above | 0 | 2 | 1 | 0 | 0
  Platelets: Missing | 1 | 0 | 1 | 0 | 1
  Monocytes: Below | 0 | 0 | 0 | 0 | 0
  Monocytes: Within | 24 | 25 | 24 | 24 | 22
  Monocytes: Above | 0 | 0 | 0 | 0 | 0
  Monocytes: Missing | 1 | 0 | 0 | 1 | 1
  Neutrophils: Below | 1 | 1 | 1 | 0 | 1
  Neutrophils: Within | 23 | 24 | 22 | 24 | 21
  Neutrophils: Above | 0 | 0 | 1 | 0 | 0
  Neutrophils: Missing | 1 | 0 | 0 | 1 | 1
  WBC: number analyzed (Participants) | 24 | 25 | 24 | 25 | 23
  WBC: Below | 1 | 1 | 1 | 0 | 1
  WBC: Within | 22 | 24 | 23 | 24 | 20
  WBC: Above | 1 | 0 | 0 | 1 | 1
  WBC: Missing | 0 | 0 | 0 | 0 | 1

24. Primary Outcome: Number of Participants With Abnormal Hematology and Biochemistry Laboratory Parameter Values at Day 31
Description: as for outcome 23
Time Frame: At Day 31
Population: The analysis was performed on the ES. Only participants for whom the specified laboratory data were available for the specified timepoint (Day 31) were included in analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | HBs-alum Group | HBs-AS03 Group | HBs-AS04 Group | HBs-AS37B Group | HBs-AS37A Group
Number analyzed (Participants) | 24 | 24 | 23 | 25 | 23
Participants
  ALT: Below | 0 | 0 | 0 | 0 | 0
  ALT: Within | 19 | 19 | 22 | 21 | 22
  ALT: Above | 5 | 5 | 1 | 3 | 1
  ALT: Missing | 0 | 0 | 0 | 1 | 0
  AST: Below | 0 | 0 | 0 | 0 | 0
  AST: Within | 22 | 23 | 21 | 24 | 23
  AST: Above | 2 | 1 | 2 | 0 | 0
  AST: Missing | 0 | 0 | 0 | 1 | 0
  Bicarbonate: Below | 0 | 0 | 0 | 0 | 0
  Bicarbonate: Within | 24 | 24 | 23 | 24 | 23
  Bicarbonate: Above | 0 | 0 | 0 | 0 | 0
  Bicarbonate: Missing | 0 | 0 | 0 | 1 | 0
  Blood urea nitrogen: Below | 0 | 0 | 0 | 0 | 0
  Blood urea nitrogen: Within | 23 | 21 | 22 | 23 | 20
  Blood urea nitrogen: Above | 1 | 3 | 1 | 1 | 3
  Blood urea nitrogen: Missing | 0 | 0 | 0 | 1 | 0
  Chloride: Below | 0 | 0 | 0 | 0 | 0
  Chloride: Within | 24 | 24 | 23 | 23 | 22
  Chloride: Above | 0 | 0 | 0 | 1 | 1
  Chloride: Missing | 0 | 0 | 0 | 1 | 0
  C Reactive Protein: Below | 0 | 0 | 0 | 0 | 0
  C Reactive Protein: Within | 22 | 23 | 17 | 25 | 20
  C Reactive Protein: Above | 2 | 1 | 6 | 0 | 3
  C Reactive Protein: Missing | 0 | 0 | 0 | 0 | 0
  Creatinine: Below | 0 | 0 | 0 | 0 | 0
  Creatinine: Within | 24 | 22 | 23 | 22 | 22
  Creatinine: Above | 0 | 2 | 0 | 2 | 1
  Creatinine: Missing | 0 | 0 | 0 | 1 | 0
  Potassium: Below | 0 | 1 | 0 | 1 | 0
  Potassium: Within | 24 | 23 | 23 | 22 | 23
  Potassium: Above | 0 | 0 | 0 | 1 | 0
  Potassium: Missing | 0 | 0 | 0 | 1 | 0
  Sodium: Below | 0 | 1 | 1 | 0 | 2
  Sodium: Within | 24 | 23 | 22 | 24 | 21
  Sodium: Above | 0 | 0 | 0 | 0 | 0
  Sodium: Missing | 0 | 0 | 0 | 1 | 0
  Eosinophils: Below | 0 | 0 | 1 | 2 | 1
  Eosinophils: Within | 23 | 23 | 22 | 21 | 22
  Eosinophils: Above | 1 | 1 | 0 | 1 | 0
  Eosinophils: Missing | 0 | 0 | 0 | 1 | 0
  Erythrocytes: Below | 0 | 1 | 5 | 1 | 2
  Erythrocytes: Within | 24 | 23 | 18 | 23 | 21
  Erythrocytes: Above | 0 | 0 | 0 | 0 | 0
  Erythrocytes: Missing | 0 | 0 | 0 | 1 | 0
  Hemoglobin: Below | 3 | 1 | 5 | 2 | 4
  Hemoglobin: Within | 21 | 23 | 17 | 22 | 19
  Hemoglobin: Above | 0 | 0 | 1 | 0 | 0
  Hemoglobin: Missing | 0 | 0 | 0 | 1 | 0
  Lymphocytes: Below | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Within | 24 | 24 | 23 | 24 | 23
  Lymphocytes: Above | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Missing | 0 | 0 | 0 | 1 | 0
  Platelets: Below | 0 | 0 | 0 | 0 | 0
  Platelets: Within | 23 | 23 | 22 | 24 | 22
  Platelets: Above | 1 | 1 | 1 | 0 | 1
  Platelets: Missing | 0 | 0 | 0 | 1 | 0
  Monocytes: Below | 1 | 0 | 0 | 0 | 0
  Monocytes: Within | 23 | 24 | 23 | 24 | 23
  Monocytes: Above | 0 | 0 | 0 | 0 | 0
  Monocytes: Missing | 0 | 0 | 0 | 1 | 0
  Neutrophils: Below | 0 | 1 | 0 | 1 | 1
  Neutrophils: Within | 24 | 23 | 23 | 23 | 20
  Neutrophils: Above | 0 | 0 | 0 | 0 | 2
  Neutrophils: Missing | 0 | 0 | 0 | 1 | 0
  WBC: Below | 1 | 1 | 0 | 1 | 1
  WBC: Within | 22 | 22 | 23 | 22 | 21
  WBC: Above | 1 | 1 | 0 | 1 | 1
  WBC: Missing | 0 | 0 | 0 | 1 | 0

25. Primary Outcome: Number of Participants With Abnormal Hematology and Biochemistry Laboratory Parameter Values at Day 38
Description: as for outcome 23
Time Frame: At Day 38
Population: The analysis was performed on the ES. Only participants for whom the specified laboratory data were available for the specified timepoint (Day 38) were included in analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | HBs-alum Group | HBs-AS03 Group | HBs-AS04 Group | HBs-AS37B Group | HBs-AS37A Group
Number analyzed (Participants) | 24 | 23 | 22 | 25 | 23
Participants
  ALT: Below | 0 | 0 | 0 | 0 | 0
  ALT: Within | 19 | 21 | 20 | 23 | 22
  ALT: Above | 4 | 2 | 2 | 2 | 1
  ALT: Missing | 1 | 0 | 0 | 0 | 0
  AST: Below | 0 | 0 | 0 | 0 | 0
  AST: Within | 22 | 22 | 22 | 24 | 23
  AST: Above | 1 | 1 | 0 | 1 | 0
  AST: Missing | 1 | 0 | 0 | 0 | 0
  Bicarbonate: Below | 1 | 0 | 1 | 0 | 1
  Bicarbonate: Within | 21 | 22 | 21 | 25 | 21
  Bicarbonate: Above | 1 | 1 | 0 | 0 | 1
  Bicarbonate: Missing | 1 | 0 | 0 | 0 | 0
  Blood urea nitrogen: Below | 0 | 0 | 0 | 0 | 0
  Blood urea nitrogen: Within | 23 | 22 | 20 | 24 | 22
  Blood urea nitrogen: Above | 0 | 1 | 2 | 1 | 1
  Blood urea nitrogen: Missing | 1 | 0 | 0 | 0 | 0
  Chloride: Below | 0 | 0 | 0 | 0 | 1
  Chloride: Within | 22 | 23 | 22 | 25 | 22
  Chloride: Above | 1 | 0 | 0 | 0 | 0
  Chloride: Missing | 1 | 0 | 0 | 0 | 0
  C Reactive Protein: Below | 0 | 0 | 0 | 0 | 0
  C Reactive Protein: Within | 19 | 20 | 17 | 24 | 21
  C Reactive Protein: Above | 4 | 3 | 5 | 1 | 2
  C Reactive Protein: Missing | 1 | 0 | 0 | 0 | 0
  Creatinine: Below | 0 | 0 | 0 | 0 | 0
  Creatinine: Within | 22 | 21 | 21 | 25 | 21
  Creatinine: Above | 1 | 2 | 1 | 0 | 2
  Creatinine: Missing | 1 | 0 | 0 | 0 | 0
  Potassium: Below | 0 | 0 | 1 | 0 | 0
  Potassium: Within | 23 | 23 | 20 | 25 | 22
  Potassium: Above | 0 | 0 | 1 | 0 | 1
  Potassium: Missing | 1 | 0 | 0 | 0 | 0
  Sodium: Below | 0 | 1 | 0 | 0 | 1
  Sodium: Within | 23 | 22 | 22 | 25 | 22
  Sodium: Above | 0 | 0 | 0 | 0 | 0
  Sodium: Missing | 1 | 0 | 0 | 0 | 0
  Eosinophils: Below | 0 | 1 | 0 | 0 | 1
  Eosinophils: Within | 21 | 21 | 22 | 24 | 22
  Eosinophils: Above | 1 | 1 | 0 | 1 | 0
  Eosinophils: Missing | 2 | 0 | 0 | 0 | 0
  Erythrocytes: Below | 1 | 0 | 1 | 1 | 1
  Erythrocytes: Within | 22 | 23 | 21 | 23 | 22
  Erythrocytes: Above | 0 | 0 | 0 | 1 | 0
  Erythrocytes: Missing | 1 | 0 | 0 | 0 | 0
  Hemoglobin: Below | 3 | 1 | 6 | 2 | 5
  Hemoglobin: Within | 20 | 22 | 16 | 23 | 18
  Hemoglobin: Above | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Missing | 1 | 0 | 0 | 0 | 0
  Lymphocytes: Below | 0 | 1 | 0 | 0 | 1
  Lymphocytes: Within | 22 | 22 | 21 | 25 | 22
  Lymphocytes: Above | 0 | 0 | 1 | 0 | 0
  Lymphocytes: Missing | 2 | 0 | 0 | 0 | 0
  Platelets: Below | 0 | 0 | 0 | 0 | 0
  Platelets: Within | 23 | 23 | 20 | 25 | 22
  Platelets: Above | 0 | 0 | 2 | 0 | 1
  Platelets: Missing | 1 | 0 | 0 | 0 | 0
  Monocytes: Below | 0 | 0 | 0 | 0 | 0
  Monocytes: Within | 22 | 23 | 21 | 25 | 23
  Monocytes: Above | 0 | 0 | 1 | 0 | 0
  Monocytes: Missing | 2 | 0 | 0 | 0 | 0
  Neutrophils: Below | 3 | 2 | 0 | 1 | 0
  Neutrophils: Within | 18 | 19 | 22 | 23 | 23
  Neutrophils: Above | 1 | 2 | 0 | 1 | 0
  Neutrophils: Missing | 2 | 0 | 0 | 0 | 0
  WBC: Below | 3 | 2 | 0 | 0 | 0
  WBC: Within | 19 | 19 | 21 | 24 | 23
  WBC: Above | 1 | 2 | 1 | 1 | 0
  WBC: Missing | 1 | 0 | 0 | 0 | 0

26. Primary Outcome: Number of Participants With Abnormal Hematology and Biochemistry Laboratory Parameter Values at Day 61
Description: as for outcome 23
Time Frame: At Day 61
Population: The analysis was performed on the ES. Only participants for whom the specified laboratory data were available for the specified timepoint (Day 61) were included in analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | HBs-alum Group | HBs-AS03 Group | HBs-AS04 Group | HBs-AS37B Group | HBs-AS37A Group
Number analyzed (Participants) | 24 | 24 | 23 | 25 | 23
Participants
  ALT: Below | 0 | 0 | 0 | 0 | 0
  ALT: Within | 21 | 20 | 21 | 23 | 20
  ALT: Above | 3 | 4 | 2 | 2 | 3
  ALT: Missing | 0 | 0 | 0 | 0 | 0
  AST: Below | 0 | 0 | 0 | 0 | 0
  AST: Within | 21 | 21 | 22 | 24 | 22
  AST: Above | 3 | 3 | 1 | 1 | 1
  AST: Missing | 0 | 0 | 0 | 0 | 0
  Bicarbonate: Below | 0 | 0 | 0 | 2 | 1
  Bicarbonate: Within | 24 | 23 | 23 | 23 | 22
  Bicarbonate: Above | 0 | 1 | 0 | 0 | 0
  Bicarbonate: Missing | 0 | 0 | 0 | 0 | 0
  Blood urea nitrogen: Below | 0 | 0 | 0 | 0 | 0
  Blood urea nitrogen: Within | 23 | 22 | 21 | 25 | 23
  Blood urea nitrogen: Above | 1 | 2 | 2 | 0 | 0
  Blood urea nitrogen: Missing | 0 | 0 | 0 | 0 | 0
  Chloride: Below | 0 | 0 | 0 | 0 | 1
  Chloride: Within | 24 | 23 | 22 | 25 | 22
  Chloride: Above | 0 | 1 | 1 | 0 | 0
  Chloride: Missing | 0 | 0 | 0 | 0 | 0
  C Reactive Protein: Below | 0 | 0 | 0 | 0 | 0
  C Reactive Protein: Within | 20 | 21 | 17 | 24 | 20
  C Reactive Protein: Above | 4 | 3 | 5 | 1 | 3
  C Reactive Protein: Missing | 0 | 0 | 1 | 0 | 0
  Creatinine: Below | 0 | 0 | 0 | 0 | 0
  Creatinine: Within | 23 | 21 | 22 | 24 | 22
  Creatinine: Above | 1 | 3 | 1 | 1 | 1
  Creatinine: Missing | 0 | 0 | 0 | 0 | 0
  Potassium: Below | 0 | 0 | 1 | 0 | 0
  Potassium: Within | 23 | 21 | 22 | 24 | 23
  Potassium: Above | 1 | 3 | 0 | 1 | 0
  Potassium: Missing | 0 | 0 | 0 | 0 | 0
  Sodium: Below | 0 | 0 | 0 | 0 | 2
  Sodium: Within | 24 | 23 | 23 | 25 | 21
  Sodium: Above | 0 | 1 | 0 | 0 | 0
  Sodium: Missing | 0 | 0 | 0 | 0 | 0
  Eosinophils: Below | 0 | 0 | 1 | 0 | 1
  Eosinophils: Within | 21 | 23 | 22 | 24 | 22
  Eosinophils: Above | 1 | 1 | 0 | 1 | 0
  Eosinophils: Missing | 2 | 0 | 0 | 0 | 0
  Erythrocytes: Below | 1 | 1 | 4 | 3 | 0
  Erythrocytes: Within | 22 | 23 | 19 | 21 | 23
  Erythrocytes: Above | 0 | 0 | 0 | 1 | 0
  Erythrocytes: Missing | 1 | 0 | 0 | 0 | 0
  Hemoglobin: Below | 4 | 1 | 5 | 4 | 3
  Hemoglobin: Within | 19 | 23 | 18 | 21 | 20
  Hemoglobin: Above | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Missing | 1 | 0 | 0 | 0 | 0
  Lymphocytes: number analyzed (Participants) | 23 | 24 | 23 | 25 | 23
  Lymphocytes: Below | 0 | 0 | 0 | 0 | 1
  Lymphocytes: Within | 23 | 24 | 23 | 25 | 22
  Lymphocytes: Above | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Missing | 0 | 0 | 0 | 0 | 0
  Platelets: Below | 0 | 0 | 0 | 0 | 0
  Platelets: Within | 22 | 22 | 21 | 24 | 23
  Platelets: Above | 0 | 2 | 2 | 0 | 0
  Platelets: Missing | 2 | 0 | 0 | 1 | 0
  Monocytes: number analyzed (Participants) | 23 | 24 | 23 | 25 | 23
  Monocytes: Below | 0 | 0 | 0 | 1 | 0
  Monocytes: Within | 23 | 24 | 23 | 24 | 23
  Monocytes: Above | 0 | 0 | 0 | 0 | 0
  Monocytes: Missing | 0 | 0 | 0 | 0 | 0
  Neutrophils: number analyzed (Participants) | 23 | 24 | 23 | 25 | 23
  Neutrophils: Below | 0 | 0 | 1 | 2 | 0
  Neutrophils: Within | 21 | 23 | 22 | 22 | 23
  Neutrophils: Above | 2 | 1 | 0 | 1 | 0
  Neutrophils: Missing | 0 | 0 | 0 | 0 | 0
  WBC: Below | 1 | 2 | 0 | 1 | 0
  WBC: Within | 20 | 21 | 23 | 22 | 22
  WBC: Above | 2 | 1 | 0 | 2 | 1
  WBC: Missing | 1 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited AEs: within 14 days after any vaccination. Unsolicited AEs: within 31 days after any vaccination. All-cause mortality, SAEs, MAEs, AEs leading to withdrawal and pIMDs: from first vaccination (Day 1) until study end (Day 361)
Arm/Group | HBs-alum Group | HBs-AS03 Group | HBs-AS04 Group | HBs-AS37B Group | HBs-AS37A Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/24 | 0/25 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/24 | 1/25 | 0/23
Other Adverse Events (participants affected / at risk) | 24/25 | 21/25 | 23/24 | 23/25 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HBs-alum Group (N=25) | HBs-AS03 Group (N=25) | HBs-AS04 Group (N=24) | HBs-AS37B Group (N=25) | HBs-AS37A Group (N=23)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HBs-alum Group (N=25) | HBs-AS03 Group (N=25) | HBs-AS04 Group (N=24) | HBs-AS37B Group (N=25) | HBs-AS37A Group (N=23)
Administration site pain (General disorders) | 7 (7) | 20 (32) | 22 (37) | 18 (30) | 21 (32)
Fatigue (General disorders) | 15 (18) | 14 (18) | 12 (18) | 14 (19) | 11 (16)
Malaise (General disorders) | 10 (14) | 7 (9) | 8 (8) | 4 (6) | 4 (4)
Chills (General disorders) | 4 (4) | 4 (4) | 0 (0) | 1 (2) | 3 (3)
Pyrexia (General disorders) | 2 (2) | 2 (3) | 1 (2) | 2 (3) | 1 (1)
Injection site inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Swelling face (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaccination site discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (10) | 11 (13) | 15 (28) | 9 (13) | 13 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5) | 3 (3) | 3 (3) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 13 (17) | 12 (17) | 10 (15) | 13 (18) | 12 (17)
Diarrhea (Gastrointestinal disorders) | 5 (6) | 4 (4) | 5 (5) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 7 (8) | 1 (1) | 5 (6) | 1 (2) | 2 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 2 (2)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal foot infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 5 (6) | 2 (2) | 1 (1) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2024-09-17): https://cdn.clinicaltrials.gov/large-docs/73/NCT05561673/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-28): https://cdn.clinicaltrials.gov/large-docs/73/NCT05561673/SAP_001.pdf